CLINICAL TRIAL: NCT03962062
Title: An Open-label Study of the Pharmacokinetics and Safety of a Single Dose of Moxidectin Per Oral in Subjects Aged 4 to 17 Years With (or at Risk of) Onchocerciasis to Identify an Optimal Dose for Treatment of Children 4 to 11 Years
Brief Title: A Pharmacokinetic and Safety Study of Moxidectin to Identify an Optimal Dose for Treatment of Children 4 to 11 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MDGH-MOX-1006
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-12

CONDITIONS: Onchocerciasis
MeSH Terms: conditions — Onchocerciasis | interventions — moxidectin

STUDY DESIGN:
Intervention Model Description: Prospective, age-stratified, adaptive, open-label, single-dose study with 3, age-defined cohorts. Cohort 1 (12 to 17 years, n = 9) and Cohort 2 (8 to 11 years, n = 9) will receive moxidectin 8 mg. Cohort 3 (4 to 7 years, n = 9) will receive moxidectin at a dose to be determined from safety and pharmacokinetic data analyses of Cohorts 1 and 2.
  If the starting dose for Cohorts 2 and 3 results in at least 3 subjects with moxidectin exposures above the target range, a revised dose will be determined in decrements of 2 mg and the Cohort(s) will be repeated with at least 9 new subjects. For Cohort 3, if the starting dose results in at least 3 subjects with moxidectin exposures below the target range, a revised dose will be determined in increments of 2 mg to a maximum dose of 8 mg.Therefore, it is expected that the study will enroll 27 subjects. However, if additional cohorts are required to meet pharmacokinetic outcomes, up to a maximum of 63 subjects may be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: 12-17 years (Experimental): Moxidectin 8mg per oral, single dose
  Interventions: Drug: Moxidectin
- Cohort 2: 8-11 years (Experimental): Moxidectin 8mg (or lower dose) per oral, single dose
  Interventions: Drug: Moxidectin
- Cohort 3: 4-7 years (Experimental): Moxidectin single dose, determined by population pharmacokinetic modelling including data from Cohorts 1 and 2
  Interventions: Drug: Moxidectin

INTERVENTIONS:
Drug: Moxidectin — 2 mg tablets

SUMMARY:
The primary purpose of this study is to determine a dose of moxidectin for children 4 to 11 years that is equivalent to an 8 mg dose administered for treatment of onchocerciasis in people 12 years and over. The secondary purpose is to evaluate the safety and pharmacokinetics of a single dose of moxidectin in children and adolescents aged 4 to 17 years.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 4 to 17 years, inclusive:

   1. Cohort I: 12 to 17 years;
   2. Cohort II: 8 to 11 years;
   3. Cohort III: 4 to 7 years;
2. Live in a region designated by the World Health Organization (WHO) as endemic for O. volvulus infection (World Health Organization, 2019). Specifically, participants will be recruited from the Kpassa sub-district of the Nkwanta North district.The specific communities will include Wii, Jagri-Do, and Azua where mass drug administration with ivermectin for onchocerciasis commenced in October 2017;
3. Willing and able to remain at the study clinic from Screening up to Day 7;
4. Provision of parental or guardian written informed consent and assent / lack of expression of 'deliberate objection' (as appropriate for age);
5. Females of childbearing potential must commit to using a reliable method of contraception as per local family planning guidelines from Baseline (pre-treatment on Day 0) until approximately 6 months after treatment with study drug.

Exclusion Criteria:

1. History of serious medical or psychiatric condition which, in the opinion of the investigator, would put the subject at increased risk by participating in the study or jeopardize study outcomes;
2. Known or suspected concurrent clinically significant renal, cardiac, pulmonary, vascular, metabolic (thyroid disorders, adrenal disease), immunological disorders or malignancy, congenital heart disease, chronic lung disease;
3. Has received an investigational product within 28 days or 5 half-lives of Baseline, whichever is longer;
4. Has received ivermectin or any other anti-helminthic treatments within 28 days of Baseline;
5. Has received a vaccination within 7 days of Baseline;
6. Known or suspected hypersensitivity to macrocyclic lactones or excipients used in the formulation of moxidectin;
7. Poor venous access;
8. Unable to swallow tablets (flat oval, 8.0 millimeters (mm) x 4.5 mm x 3.0 mm);
9. Weight:

   1. Cohort I (12 to 17 years): < 30 kg;
   2. Cohort II (8 to 11 years): < 18 kg;
   3. Cohort III (4 to 7 years): < 12 kg;
10. Clinically relevant laboratory abnormalities at Screening, including:

    1. Hemoglobin < 9.5 grams per deciliter (g/dL);
    2. Neutrophil (granulocyte) count < 1.5 x 109/L;
    3. Platelet count < 110 x 109/L;
    4. Alanine aminotransferase (ALT) > 1.5 times the upper limit of normal range (ULN);
    5. Total bilirubin > 1.5 times ULN;
11. Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV) positive;
12. Known or suspected malaria or other ongoing viral, bacterial, or plasmodium infection at Screening and/or Baseline;
13. Loa loa co-infection;
14. Unwilling, unlikely or unable to comply with all protocol specified assessments;
15. For females of child bearing potential, pregnant or breastfeeding, or planning to become pregnant;
16. Previous enrolment in this study;
17. Is a sibling of another child already enrolled in this study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas O Opoku, MD, Principal Investigator — University of Health and Allied Sciences School of Public Health, Hohoe, Ghana
Locations (1):
- University of Health and Allied Services School of Public Health, Hohoe, Volta Region, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data in the form of data listings and SDTM and ADaM datasets may be available for sharing on application to the Sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available 12 months after publication.
Access Criteria: Provision of a methodologically sound and relevant proposal detailing the intended use of the data and relevant ethics approval for the proposed analysis, as applicable.

REFERENCES:
- [Result] Opoku NO, Doe F, Agbogah ME, Laryea R, Gordor SK, Donkor BS, Anyomitse E, Kugali D, van Zutphen-van Geffen M, Navarro DJ, Rayner CR, Patel K, Kuesel AC, Lowe M, Kinrade S. Identification of a moxidectin dose for 4- to 11-year-old children to support registration and potential use for onchocerciasis elimination: results of an open-label pharmacokinetic and safety study. Parasit Vectors. 2025 Jul 24;18(1):295. doi: 10.1186/s13071-025-06891-z. PMID 40707999
- See also: Identification of a moxidectin dose for 4- to 11-year-old children to support registration and potential use for onchocerciasis elimination: results of an open-label pharmacokinetic and safety study. — https://parasitesandvectors.biomedcentral.com/articles/10.1186/s13071-025-06891-z

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was screened on 29 March 2021 and the last participant last study visit was completed on 28 September 2022. Participants were recruited from communities in the Kpassa sub-district of the Oti region in Ghana, which is endemic for onchocerciasis.
Groups:
- 12 to 17 Years MOX 8 mg: Cohort 1: Nine (9) participants aged 12 to 17 years at Screening received a single oral dose of moxidectin 8 mg and were followed for 24 weeks for pharmacokinetic and safety outcomes.
- 8 to 11 Years MOX 8 mg: Cohort 2: Nine (9) participants aged 8 to 11 years at Screening received a single oral dose of moxidectin 8 mg and were followed for 24 weeks for pharmacokinetic and safety outcomes.
- 8 to 11 Years MOX 6 mg: Cohort 2: Nine (9) participants aged 8 to 11 years at Screening received a single oral dose of moxidectin 6 mg and were followed for 24 weeks for pharmacokinetic and safety outcomes.
- 4 to 7 Years MOX 4 mg: Cohort 3: Nine (9) participants aged 4 to 7 years at Screening received a single oral dose of moxidectin 4 mg and were followed for 24 weeks for pharmacokinetic and safety outcomes.
Period: Overall Study
Arm/Group | 12 to 17 Years MOX 8 mg | 8 to 11 Years MOX 8 mg | 8 to 11 Years MOX 6 mg | 4 to 7 Years MOX 4 mg
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and Baseline characteristics were analyzed in the Safety Analysis Set, which included all participants who provided signed informed consent/ assent and whose eligibility was confirmed on Day 0, and the Pharmacokinetic Analysis Set, which included all participants who received moxidectin and provided a minimum number of plasma samples for the determination of PK parameters. As no subjects were excluded from any analysis set, the data within these data sets is identical.
Groups:
- 12 to 17 Years Moxidectin 8 mg: Cohort 1: Nine (9) participants aged 12 to 17 years at Screening received a single oral dose of moxidectin 8 mg and were followed for 24 weeks for pharmacokinetic and safety outcomes.
- 8 to 11 Years Moxidectin 6 mg: Cohort 2: Nine (9) participants aged 8 to 11 years at Screening received a single oral dose of moxidectin 6 mg and were followed for 24 weeks for pharmacokinetic and safety outcomes.
- 8 to 11 Years Moxidectin 8 mg: Cohort 2: Nine (9) participants aged 8 to 11 years at Screening received a single oral dose of moxidectin 8 mg and were followed for 24 weeks for pharmacokinetic and safety outcomes.
- 4 to 7 Years Moxidectin 4 mg: Cohort 3: Nine (9) participants aged 4 to 7 years at Screening received a single oral dose of moxidectin 4 mg and were followed for 24 weeks for pharmacokinetic and safety outcomes.
- Total: Total of all reporting groups
Arm/Group | 12 to 17 Years Moxidectin 8 mg | 8 to 11 Years Moxidectin 6 mg | 8 to 11 Years Moxidectin 8 mg | 4 to 7 Years Moxidectin 4 mg | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (1.66) | 9.1 (1.05) | 9.7 (0.87) | 5.4 (1.33) | 9.5 (3.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 5 | 6 | 21
  Male | 5 | 3 | 4 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 9 | 9 | 36
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Ghana | 9 | 9 | 9 | 9 | 36
Height [Mean (Standard Deviation); unit: cm] | 149.74 (10.318) | 130.09 (9.307) | 133.11 (10.590) | 108.81 (7.922) | 130.44 (17.381)
Weight [Mean (Standard Deviation); unit: kg] | 39.42 (8.754) | 25.89 (4.567) | 27.13 (4.844) | 16.90 (2.662) | 27.34 (9.766)
BMI [Mean (Standard Deviation); unit: kg/m2] | 17.39 (1.745) | 15.19 (1.068) | 15.23 (1.120) | 14.20 (0.919) | 15.50 (1.683)
Mean upper arm circumference at Screening [Mean (Standard Deviation); unit: cm] | 21.78 (2.065) | 18.42 (0.981) | 18.66 (1.591) | 15.68 (1.347) | 18.63 (2.644)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve of Moxidectin.
Description: Moxidectin concentration in plasma collected at pre-specified intervals after dosing with oral moxidectin determined using a validated liquid chromatography-mass spectrometry(MS)/MS method.
Time Frame: Pre-dose (Screening) and post-dose at Hours 1, 2, 4, 8, 24 and 72 and Days 7, 14 and 28.
Population: The Pharmacokinetic Analysis Set included all participants who received moxidectin and provided a minimum number of plasma samples for the determination of Pharmacokinetic (PK) parameters, defined as one (1) sample taken at each of hours 4, 24 and 72, plus one (1) sample taken at either Day 14 or Day 28. Subjects were analyzed according to the dose received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hr*ng/mL)/mg
Arm/Group | 12 to 17 Years MOX 8 mg | 8 to 11 Years MOX 6 mg | 8 to 11 Years MOX 8 mg | 4 to 7 Years MOX 4 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
(hr*ng/mL)/mg | 2680 (24.7) | 2230 (52.3) | 3310 (23.0) | 1880 (26.5)

2. Secondary Outcome: Area Under the Concentration Versus Time Curve (Zero to Infinity) of Moxidectin
Description: as for outcome 1
Time Frame: Pre-dose (Screening) and post-dose at Hours 1, 2, 4, 8, 24 and 72, Days 7, 14 and 28 and Week 12.
Population: The Pharmacokinetic Analysis Set included all participants who received moxidectin and provided a minimum number of plasma samples for the determination of PK parameters, defined as one (1) sample taken at each of hours 4, 24 and 72, plus one (1) sample taken at either Day 14 or Day 28. Subjects were analyzed according to the dose received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hr*ng/mL)/mg
Arm/Group | 12 to 17 Years MOX 8 mg | 8 to 11 Years MOX 6 mg | 8 to 11 Years MOX 8 mg | 4 to 7 Years MOX 4 mg
Number analyzed (Participants) | 8 | 9 | 9 | 9
(hr*ng/mL)/mg | 3140 (24.8) | 2490 (59.2) | 3780 (29.2) | 2000 (29.3)

3. Secondary Outcome: Maximum Observed Plasma Concentrations (Cmax) of Moxidectin
Description: as for outcome 1
Time Frame: Pre-dose (Screening) and post-dose at Hours 1, 2, 4 and 8.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 12 to 17 Years MOX 8 mg | 8 to 11 Years MOX 6 mg | 8 to 11 Years MOX 8 mg | 4 to 7 Years MOX 4 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
ng/mL | 83.1 (19.1) | 82.1 (41.2) | 115 (25.6) | 86.4 (28.3)

4. Secondary Outcome: Incidence and Severity of Adverse Events.
Description: Incidence and severity of adverse events, assessed by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Paediatric Adverse Events, Version 2.1.
Time Frame: Day 0 to Week 24 inclusive.
Population: The Safety Analysis Set included all participants who received any exposure to moxidectin. Subjects were analyzed according to the dose received.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 to 17 Years MOX 8 mg | 8 to 11 Years MOX 6 mg | 8 to 11 Years MOX 8 mg | 4 to 7 Years MOX 4 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  All Treatment-emergent Adverse Events (TEAEs) | 4 | 7 | 6 | 7
  TEAEs by Severity Grade 1 Mild | 3 | 6 | 6 | 6
  Grade 2 Moderate | 1 | 1 | 1 | 2
  Grade 3 Severe | 0 | 0 | 0 | 1
  Grade 4 Life-threatening | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 to 24 weeks.
Groups:
- Overall: Combined Cohorts 1 to 3: 36 participants
Arm/Group | 12 to 17 Years MOX 8 mg | 8 to 11 Years MOX 6 mg | 8 to 11 Years MOX 8 mg | 4 to 7 Years MOX 4 mg | Overall
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/36
Other Adverse Events (participants affected / at risk) | 4/9 | 7/9 | 6/9 | 7/9 | 24/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 to 17 Years MOX 8 mg (N=9) | 8 to 11 Years MOX 6 mg (N=9) | 8 to 11 Years MOX 8 mg (N=9) | 4 to 7 Years MOX 4 mg (N=9) | Overall (N=36)
Malaria (Infections and infestations) | 1 (1) | 5 (7) | 4 (6) | 4 (6) | 14 (20)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hookworm infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
False positive investigation result (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT03962062/Prot_SAP_ICF_001.pdf